CLINICAL TRIAL: NCT05546684
Title: The Effect of Foot Bath on Postoperative Sleep Quality in Patients Undergoing Transurethral Resection: A Randomized Controlled Study
Brief Title: The Effect of Foot Bath on Postoperative Sleep Quality in Patients Undergoing Transurethral Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Figen Dıgın, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TUTF-GOBAEK 2022/152
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: The Effect of Footbath
Keywords: foot bath, sleep quality,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot bath (Experimental): Individuals who apply to the urology service for TURP or TURM will be informed about the study 1 day before the surgery, and the questions in the patient introduction form will be asked to the patients who declared that they agreed to participate in the study in written and verbal form. On the morning of the surgery, the RCSQ will be applied to the patients to determine the preoperative sleep quality, and the Patient follow-up form will be applied to determine the confounding factors that may affect the sleep. The patient's feet will be kept in the footbath device for ten minutes. After the foot bath, the patient's feet will be completely dried with a towel and the existing socks and anti-embolic socks will be put on again. On the morning of the 1st postoperative day, the patient will be asked the questions in the RCSQ and the follow-up form, and the data collection process of the study will be terminated.
  Interventions: Other: footbath
- Control Group (No Intervention): After informing the individuals who applied to the urology service for TURP or TURM about the study, the researcher will receive their informed consent in written form. The information required for the study of the patients in the control group 1 day before the operation will be recorded in the Patient Information Form by the service nurse. On the morning of the surgery, the RCSQ will be applied to the patients to determine the preoperative sleep quality and the Patient follow-up form will be applied to determine the confounding factors that may affect sleep. In the morning of the first day after the surgery, the RCSQ will be applied to the patients to determine the sleep quality on the postoperative day 0, and the Patient follow-up form will be applied to determine other possible factors that may affect sleep, and the data collection process of the study will be terminated. No foot bath application will be in question for the patients in the control group.

INTERVENTIONS:
Other: footbath — footbath for patients before sleeping
  Arms: foot bath

SUMMARY:
Of the patients who meet the inclusion criteria, 82 will be determined prospectively. Randomization will be determined by means of a computer program called Research randomiser, provided that the number of patients in the experimental and control groups is equal (41:41), regardless of the characteristics of the patients such as age and gender. The group to which foot bath will be applied will be the experimental group. Other patients will be included in the control group.

Patients who do not meet the study criteria and do not agree to participate in the random selection will not be included in the study.

Experimental group: Individuals who applied to the urology service for TURP or TURM will be informed about the study 1 day before the operation, and the questions in the patient introduction form will be asked to the patients who declared that they agreed to participate in the study in writing and verbally. RCSQ to determine preoperative sleep quality for patients on the morning of surgery and Patient Methods to be applied / Research protocol to identify confounding factors that may affect sleep (Fill in the appropriate section below).

Eligibility assessment: Of the patients who meet the inclusion criteria, 82 will be determined prospectively.

Providing randomization and separation for intervention: Randomization will be determined by means of a computer program called Research randomiser, provided that the number of patients in the experimental and control groups is equal (41:41), regardless of the characteristics of the patients, such as age and gender. The group to which foot bath will be applied will be the experimental group. Other patients will be included in the control group.

Patients who do not meet the study criteria and do not agree to participate in the random selection will not be included in the study.

Experimental group: Individuals who applied to the urology service for TURP or TURM will be informed about the study 1 day before the operation, and the questions in the patient introduction form will be asked to the patients who declared that they agreed to participate in the study in writing and verbally. On the morning of the surgery, the RCSQ will be applied to the patients to determine the preoperative sleep quality and the Patient follow-up form will be applied to determine the confounding factors that may affect sleep, and after the patient comes from the surgery and the sedation effects have passed, at 21:00 (to prevent the patient from doing any activity after the application and to rest after the foot bath). It was determined as 21:00-22:00 hours for the purpose.) socks, etc., if any, on both feet of the patient. clothes will be removed. In case of using antiembolic stockings, the patient's stockings will be rolled up to the ankle for footbath application (with the approval of the physician). The foot will be examined visually and with the hands and it will be determined that it does not show any signs of disease (pressure injury, discoloration, wound, etc.). The patient will be informed that the footbath device is disinfected before each use and that water-proof bags will be placed on the device to prevent the foot and water from coming into contact with the device in order to allow repeated use. The temperature of the water will be adjusted to 400C with an infrared temperature meter (Non-contact digital thermometer) and both feet will be placed inside the footbath device. The patient's feet will be kept in the footbath device for ten minutes. After the foot bath, the patient's feet will be completely dried with a towel and the existing socks and anti-embolic socks will be put on again (Meltem Nurse). On the morning of the first postoperative day, the patient will be asked the questions in the RCSQ and follow-up form, and the data collection process of the study will be terminated.

Control group: After informing the individuals who applied to the urology service for TURP or TURM about the study, the researcher will receive their informed consent in written form. The information required for the study of the patients in the control group 1 day before the operation will be recorded in the Patient Information Form by the service nurse (Meltem Nurse / Gizem Nurse). On the morning of the surgery, the RCSQ will be applied to the patients to determine the preoperative sleep quality and the Patient follow-up form will be applied to determine the confounding factors that may affect sleep. In the morning of the first day after the surgery, the RCSQ will be applied to the patients to determine the sleep quality on the postoperative day 0 and the Patient follow-up form will be applied to determine other possible factors that may affect sleep, and the data collection process of the study will be terminated. No foot bath application will be in question for the patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily agreed to participate in the study, accepted random selection, were adults, did not have visual/verbal/auditory communication difficulties and mental disabilities that prevented them from answering the questions in the scale, were applied TURP or TURM.

Exclusion Criteria:

* Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
sleep quality | 1 year
  The Richards-Campbell Sleep Questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Dığın, Dr, Study Chair — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)